CLINICAL TRIAL: NCT01305603
Title: Dual TAP Block Characteristics - Evaluation of Local Anesthetic Distribution by MR Scanning
Brief Title: Ultrasound-guided Dual TAP Block: Magnetic Resonance (MR) Evaluation of the Distribution of Local Anesthetic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Jens Borglum Neimann, Jens Børglum Neimann, MD, PhD, MBA, Consultant Anesthetist, Bispebjerg Hospital, Copenhagen University Hospital, Department of Anesthesia and Intensive Care Medicine, Bispebjerg Bakke 23, DK-2400 Copenhagen NV, Denmark, Bispebjerg Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: BBH-USG-PNB-1
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Anesthetics, Local; Injections; Nerve Block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dual TAP block (Active Comparator): Dual TAP block on one side on the abdomen. Classical (or single) TAP on the contra lateral side of the abdomen; supplemented with a sham injection to ensure double blindness.
  Interventions: Drug: Bupivacaine; Procedure: Injection
- Classical (or single) TAP block (Active Comparator): Dual TAP block on one side on the abdomen. Classical (or single) TAP on the contra lateral side of the abdomen; supplemented with a sham injection to ensure double blindness
  Interventions: Drug: Bupivacaine; Procedure: Injection

INTERVENTIONS:
Drug: Bupivacaine — On both sides of the abdomen 30 ml of bupivacaine 2.5 mg/ml will be injected. This is a total of 60 ml of bupivacaine 2.5 mg/ml.
  Other Names: Local anesthetic
Procedure: Injection — Injection under ultrasound-guidance
  Other Names: Nerve blocks

SUMMARY:
Using Magnetic resonance (MR) scanning and ultrasonography the investigators wish to investigate, in what way a known volume of local anesthetic injectate will be distributed in the transverse abdominis plane (TAP) in young healthy male volunteers. The investigators compare the anatomical distribution of the local anesthetic injectate in the TAP when performing an ultrasound-guided classical TAP block and a Dual TAP block. The investigators also want to compare the spread of anesthetized frontal dermatomes when performing an ultrasound-guided classical TAP block and a Dual TAP block.

DETAILED DESCRIPTION:
There has been much debate as to what extent the classical TAP block will anesthetize more than the frontal dermatomes (TH10-Th12/L1). Some cadaver studies have been performed with injection of dye in the classical TAP. However, it is still not clear whether a single injection of local anesthetic in the classical TAP block position will reach the more cephalad and medial intercostal TAP plexus (Th6-Th9). In this study the investigators use MR scanning and ultrasonography to investigate in what way a known volume of local anesthetic injectate will be distributed in the transverse abdominis plane (TAP) in young healthy male volunteers. The investigators compare the anatomical distribution of the local anesthetic injectate in the TAP when performing an ultrasound-guided classical TAP block and a Dual TAP block. The investigators also want to compare the spread of anesthetized frontal dermatomes when performing an ultrasound-guided classical TAP block and a Dual TAP block.

ELIGIBILITY:
Inclusion Criteria:

* healthy male
* 18 years old or more
* had no previous abdominal surgery
* no regular medication
* no coagulation disorders
* no claustrophobia

Exclusion Criteria:

* if the volunteer is not able to accept an uncomplicated administration of a classical (single) or dual TAP block

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Distribution of local anesthetic evaluated by MR scanning | 30 minutes after administering the TAP blocks

SECONDARY OUTCOMES:
Spread of anesthetized frontal dermatomes | 30 minutes after administering the TAP blocks

CONTACTS AND LOCATIONS:
Overall Officials: Jens B Neimann, MD, PhD, MBA, Principal Investigator — Dept. of Anesthesia, Bispebjerg Hospital, Copenhagen University Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen University Hospital, Copenhagen, Capital Region of Denmark, Denmark

REFERENCES:
- [Background] Petersen PL, Mathiesen O, Torup H, Dahl JB. The transversus abdominis plane block: a valuable option for postoperative analgesia? A topical review. Acta Anaesthesiol Scand. 2010 May;54(5):529-35. doi: 10.1111/j.1399-6576.2010.02215.x. Epub 2010 Feb 17. PMID 20175754